CLINICAL TRIAL: NCT00370799
Title: A Randomized, Prospective, Double-Blind Controlled Evaluation of the Effectiveness of Caudal Epidural Injections in Lumbar Disc Herniations, Spinal Stenosis, Discogenic Pain, and Post-Lumbar Laminectomy Syndrome
Brief Title: Effectiveness of Caudal Epidural Injections in Treatment of Chronic Low Back and Lower Extremity Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: protocol 10
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Low Back Pain
Keywords: Caudal Epidural injections; lumbar disc herniation; spinal stenosis; discogenic pain; post-lumbar laminectomy syndrome
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement; Spinal Stenosis | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- local anesthetic (Active Comparator): Group 1. local anesthetics only
  Interventions: Drug: Caudal epidural injection
- Local anesthetic with generic Celestone (Active Comparator): Group 2. local anesthetic with 6mg of non-particulate Celestone
  Interventions: Drug: Caudal Epidural Injection with generic Celestone
- Local anesthetic with Celestone (Active Comparator): Group 3. local anesthetic with 6 mg of brand nameCelestone
  Interventions: Drug: Caudal Epidural Injection with Celestone
- Local anesthetic with DepoMedrol (Active Comparator): Group 4. local anesthetic with 40 mg of alcohol-free DepoMedrol
  Interventions: Drug: Caudal Epidural Injection with DepoMedrol

INTERVENTIONS:
Drug: Caudal epidural injection — group 1: Caudal epidural injection local anesthetics only
  Other Names: Group 1
  Arms: local anesthetic
Drug: Caudal Epidural Injection with generic Celestone — Group 2. Caudal Epidural Injection local anesthetic with 6mg of non-particulate Celestone
  Other Names: Group 2
  Arms: Local anesthetic with generic Celestone
Drug: Caudal Epidural Injection with Celestone — Group 3. Caudal Epidural Injection with local anesthetic with 6 mg of brand name Celestone
  Other Names: Group 3
  Arms: Local anesthetic with Celestone
Drug: Caudal Epidural Injection with DepoMedrol — Group 4. local anesthetic with 40 mg of alcohol-free DepoMedrol
  Other Names: Group 4
  Arms: Local anesthetic with DepoMedrol

SUMMARY:
To demonstrate clinically significant improvements or lack thereof in the caudal epidural patients with our without steroids.

To evaluate differences in outcomes in patients receiving steroids compared to those patients randomized to the local anesthetic group who did not receive steroids.

To assess improvements among patients and compare steroid groups with each other and local anesthetic group.

To evaluate and compare the adverse event profile in all patients

DETAILED DESCRIPTION:
Patients with chronic low back pain of at least 6 months duration, non-responsive to conservative management with NSAIDS, physical therapy or chiropractic treatment exercises.

A single-center, prospective, controlled, double blinded, randomized study of patients in 4 groups.

* Group 1. local anesthetics only
* Group 2. local anesthetic with 6mg of non-particulate Celestone
* Group 3. local anesthetic with 6 mg of brand name Celestone
* Group 4. local anesthetic with 40 mg of alcohol-free DepoMedrol

All patients will be unblinded in 12 months.

Non-responsive patients will be unblinded after 3 months and will be crossed over to a different group

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* History of chronic, function-limiting low back pain of at least 6 months duration
* Able to give voluntary, written informed consent to participate,
* Able to understand the investigation, cooperate with the procedures, and willing to return for follow-up
* No recent surgical procedures within last three months

Exclusion Criteria:

* Cauda Equina symptoms and/or compressive radiculopathy
* Narcotic use of no greater than 100mg/day hydrocodone, 60mg Methadone. or 100mg morphine
* Uncontrolled major Depression or uncontrolled psychiatric disorder
* Uncontrolled or acute medical illnesses
* Chronic severe conditions that could interfere with outcome assessments
* Women who are pregnant or lactating
* Subjects who have participated in a clinical study with an investigational product within 30 days of enrollment
* Patients with multiple complaints involving concomitant hip osteoarthritis
* Inability to achieve proper positioning and inability to understand informed consent and protocol
* History of adverse reaction to local anesthetic or anti-inflammatory drugs and history of gastrointestinal bleeding or ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To evaluate for differences between the patients in various groups in the physical function and pain at 1, 3, 6, and 12 months post treatment | 1,3,6,12 months

SECONDARY OUTCOMES:
To assess adverse events in all four groups. | 1,3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States

REFERENCES:
- [Derived] Manchikanti L, Singh V, Cash KA, Pampati V, Damron KS, Boswell MV. Effect of fluoroscopically guided caudal epidural steroid or local anesthetic injections in the treatment of lumbar disc herniation and radiculitis: a randomized, controlled, double blind trial with a two-year follow-up. Pain Physician. 2012 Jul-Aug;15(4):273-86. PMID 22828681
- [Derived] Manchikanti L, Cash KA, McManus CD, Pampati V, Smith HS. One-year results of a randomized, double-blind, active controlled trial of fluoroscopic caudal epidural injections with or without steroids in managing chronic discogenic low back pain without disc herniation or radiculitis. Pain Physician. 2011 Jan-Feb;14(1):25-36. PMID 21267039
- [Derived] Manchikanti L, Singh V, Cash KA, Pampati V, Datta S. Management of pain of post lumbar surgery syndrome: one-year results of a randomized, double-blind, active controlled trial of fluoroscopic caudal epidural injections. Pain Physician. 2010 Nov-Dec;13(6):509-21. PMID 21102963